CLINICAL TRIAL: NCT06419608
Title: A Phase 2 Multicenter, Randomized, Double-blind, Placebo-controlled, Study to Evaluate the Efficacy and Safety of BHV-7000 Monotherapy in Major Depressive Disorder
Brief Title: Efficacy and Safety Study of BHV-7000 Monotherapy in Major Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biohaven Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Organization: Biohaven Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV7000-305
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder
Keywords: depression; depressed; depressive disorder; major depression; major depressive episode; antidepressant
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Consciousness Disorders; Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BHV-7000 (Experimental)
  Interventions: Drug: BHV-7000
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BHV-7000 — BHV-7000 75 mg taken once daily for 6 weeks
  Arms: BHV-7000
Drug: Placebo — Matching placebo taken once daily for 6 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of BHV-7000 in participants with Major Depressive Disorder (MDD)

ELIGIBILITY:
Key Inclusion Criteria:

1. Subjects experiencing a moderate to severe episode of depression.
2. Subjects experiencing a current episode of depression for at least 2 months.
3. Subjects must be willing to discontinue all psychotropic medications (other medications to treat depression) before entering the study.
4. Male and Female participants 18 to 75 years of age at the time of consent.
5. Body Mass Index (BMI) must be ≥ 18 kg/m2 and ≤ 35 kg/m2.

Key Exclusion Criteria:

1. Subjects taking more than 2 medications (other than benzodiazepines and medications targeting insomnia) to treat depression at the screening visit.
2. Subjects with a history of bipolar disorder, schizophrenia, or other neuropsychiatric conditions that may interfere with the conduct of the study.
3. Subjects with a history of medical conditions that may interfere with the conduct of the study.
4. Females who are pregnant, breastfeeding or planning to become pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Change in Montgomery- Åsberg Depression Rating Scale (MADRS) total score from baseline to week 6 | Baseline to Week 6
  The MADRS is a clinician- rated scale to assess depressive symptoms which consists of 10 items. Each item is scored on 7-point scale (0 [absence of symptoms] to 6 [severe]). A higher score represents a higher severity of the level of depression (total scores range from 0 to 60).

SECONDARY OUTCOMES:
Change in Clinical Global Clinical Impression - Severity Scale (CGI-S) total score | Baseline to Week 6
  The CGI-S is a clinician-rated scale to assess disease severity. The scale is scored on 8-point scale (0 [not assessed] to 7 [severe]). A higher score represents a higher severity illness.
Change in Snaith-Hamilton Pleasure Scale (SHAPS) total score from baseline to week 6 | Baseline to Week 6
  The SHAPS is a subject self- administered scale to measure hedonic capacity which consists of 14 items (total scores range from 0 to 14). Each item has a set of 4 possible responses (Strongly or Definitely Agree, Agree, Disagree and Strongly Disagree). A total score is derived by summing the responses to each item. A higher score represents a higher level of anhedonia.
Change in Montgomery- Åsberg Depression Rating Scale (MADRS) total score from baseline to week 1 | Baseline to Week 1
  The MADRS is a clinician- rated scale to assess depressive symptoms which consists of 10 items. Each item is scored on 7-point scale (0 [absence of symptoms] to 6 [severe]). A higher score represents a higher severity of the level of depression (total scores range from 0 to 60).
Change in Snaith-Hamilton Pleasure Scale (SHAPS) total score from baseline to week 1 | Baseline to Week 1
  The SHAPS is a subject self- administered scale to measure hedonic capacity which consists of 14 items (total scores range from 0 to 14). Each item has a set of 4 possible responses (Strongly or Definitely Agree, Agree, Disagree and Strongly Disagree). A total score is derived by summing the responses to each item. A higher score represents a higher level of anhedonia.
Change in Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q- LES-Q-SF) total score | Baseline to Week 6
  The Q-LES-Q-SF is a participant self-administered scale to assess the degree of enjoyment and satisfaction experienced in various areas of daily functioning. The form consists of 16 items. Each item is scored on 5-point scale. A higher score represents a higher level of satisfaction and enjoyment (total scores range from 14 to 70).
Number of Participants With Serious AEs (SAEs), AEs Leading to Study Drug Discontinuation, and AEs judged to be related to study medication | Screening through Week 8
  Safety and tolerability of BHV-7000 as assessed by frequency of unique subjects with SAEs; AEs leading to discontinuation; AEs judged to be related to study medication
Number of Participants With Clinically Significant Laboratory Abnormalities | Screening through Week 8
  To assess the safety and tolerability of BHV-7000. This objective will be measured by assessing the number of unique subjects with grade 3 or 4 laboratory abnormalities.
Number of Participants With Vital Sign Abnormalities | Screening through Week 8
Number of Participants With Electrocardiogram (ECG) Abnormalities specific to QTc elevation | Screening through Week 8

CONTACTS AND LOCATIONS:
Locations (62):
- United States (62):
  - IMA Clinical Research, Phoenix, Arizona
  - Pillar Clinical Research, LLC, Little Rock, Arkansas
  - WIRG, Little Rock, Arkansas
  - WRN, Rogers, Arkansas
  - Advanced Research Center, Inc., Anaheim, California
  - CIT LA, Bellflower, California
  - IPMG, Chino, California
  - WR-PRI Encino, Encino, California
  - Collaborative Neuroscience Research, LLC (CenExel - CNS), Garden Grove, California
  - CalNeuro Research Group, Los Angeles, California
  - Excell Research, Inc., Oceanside, California
  - NRC Research Institute, Orange, California
  - Anderson Clinical Research, Redlands, California
  - CIT IE, Riverside, California
  - Lumos Clinical Research Center, San Jose, California
  - Stanford, Stanford, California
  - Cenexel CNS, Torrance, California
  - Pacific Clinical Research Management Group, Upland, California
  - Sunwise Clinical Research, Walnut Creek, California
  - MCB Clinical Research Centers, Colorado Springs, Colorado
  - UConn Health, Farmington, Connecticut
  - Optum Behavioral Care of Connecticut, PC dba Comprehensive Psychiatric Care of Connecticut, Norwich, Connecticut
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Floridian Neuroscience Institute, Miami Lakes, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - K2 Medical Research, Tampa, Florida
  - Neuroscience Research Institute, West Palm Beach, Florida
  - CenExel iResearch, LLC, Decatur, Georgia
  - CenExel iResearch, LLC, Savannah, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - Revive Research Institute, Inc., Elgin, Illinois
  - Collective Medical Research, Overland Park, Kansas
  - Delricht Research, New Orleans, Louisiana
  - Headlands Pharmasite, Baltimore, Maryland
  - CBH Health, Gaithersburg, Maryland
  - Copley Clinical, Boston, Massachusetts
  - Boston Clinical Trials, Boston, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - Precise Clinical Research, Flowood, Mississippi
  - Arch Clinical Trials, St Louis, Missouri
  - IMA Clinical Research, Las Vegas, Nevada
  - Bio Behavioral Health, Toms River, New Jersey
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Neurobehavioral Research, Inc, Cedarhurst, New York
  - Bioscience Research LLC, Mount Kisco, New York
  - Berman Clinical, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - RBA, Staten Island, New York
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Scranton Medical Institute, Moosic, Pennsylvania
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Donald J. Garcia, MD, PA dba Austin Clinical Trial Partners, Austin, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Relaro Medical Trials, LLC, Dallas, Texas
  - InSite Clinical Research, LLC, DeSoto, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Aim Trials, Plano, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Alpine Reseach Organization, Clinton, Utah
  - Northwest Clinical Research Center, Bellevue, Washington